CLINICAL TRIAL: NCT05699421
Title: Universal Screening Program for Cytomegalovirus Infection in the First Trimester of Pregnancy: A Multicentre Pilot Study in the Area of Barcelona (CITEMB Study)
Brief Title: Universal Screening Program for Cytomegalovirus Infection in the First Trimester of Pregnancy (CITEMB Study)
Acronym: CITEMB
Status: Completed | Type: Observational
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Vall d'Hebron Barcelona Hospital Campus (Unknown); Hospital Clínic Sede Maternitat (Other); Germans Trias i Pujol Hospital (Other); ASSIRs Barcelona (Unknown); ASSIRs Metropolitana Nord (Unknown)
Responsible Party: Sponsor
Other Study IDs: 22/097-P
Record Dates: First submitted 2023-01-09; First posted 2023-01-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Screening
Keywords: universal screening; pregnancy; cytomegalovirus; vertical transmission; child health prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CITEMB project participants: This is a single cohort, observational prospective multicenter study. The participating centers of the Barcelona Northern Metropolitan Area are primary attention centers - ASSIR Muntanya, ASSIR Esquerra, ASSIR Santa Coloma de Gramenet, ASSIR Badalona-Sant Adrià and hospitals - Vall d'Hebron University Hospital in Barcelona, BCNatal, Hospital Clínic /Hospital Sant Joan de Déu University of Barcelona and Trias i Pujol University Hospital.
  Interventions: Other: screening programme

INTERVENTIONS:
Other: screening programme — CMV screening during the first trimester of pregnancy and neonatal

SUMMARY:
The aim of this study is to evaluate a universal cCMV screening programme in the first trimester of pregnancy in primary care in Catalonia (Spain).

DETAILED DESCRIPTION:
This is the pilot study of implementation of the CMV universal screening program in the first trimester of pregnancy Barcelona and its metropolitan area.

General objective The aim of this study is to evaluate a universal CMV screening programme in the first trimester of pregnancy in primary care.

Specific aims of this pilot study:

1. Estimate the percentage of acceptance of CMV screening in the population
2. To observe and to determine the rate of CMV primary infection in the first trimester of pregnancy
3. To identify and describe the rate of the vertical fetal infection detected through the amniocentesis of the 2nd trimester
4. To identify and describe the rate of fetal sequelae (due to the primary CMV infection in the first trimester), obtained by imaging techniques (ultrasound and MRI)
5. To identify and describe the rate of neonatal infection (congenital CMV)
6. To identify and describe the rate of sequelae for congenital CMV at one year of the child's age
7. To identify and describe the percentage rate of TOP following the diagnosis of primary infection on CMV
8. To identify and describe the rate of legal of TOP following the diagnosis of fetal infection
9. To identify and describe the rate of TOP following the diagnosis of fetal anomalies
10. To obtain and describe the annual cost of CMV screening in the first quarter in Catalonia (Spain).

ELIGIBILITY:
Inclusion Criteria:

* maternal age 16 years or older, and
* gestational age less than 14 weeks.

Exclusion Criteria:

* language barrier preventing informed consent,
* gestational age at blood sampling above 14 weeks, and
* consent withdrawal

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: women > 16 years old (reproductive age), during first trimester of pregnancy
Sampling Method: Probability Sample
Enrollment: 3357 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
CMV seroprevalence in first trimester of pregnancy | 18-19 months
  Nº IgG positive with negative IgM + IgG positive with positive IgM and high avidity) / Nº of serologies performed.
Prevalence of CMV primary infection in the first trimester of pregnancy or in the periconceptional period | 18-19 months
  Nº IgG positive with IgM positive and low or intermediate avidity / Nº serologies performed.
Fetal infection rate at 2nd trimester amniocentesis | 3-24 months
  Nº positive PCR-CMV in amniotic fluid/total amniocentesis.
Rate of fetal compromise by imaging techniques (ultrasound and MRI) after first trimester / periconceptional CMV infection | 3-24 months
  ultrasound or MRI abnormalities attributable to CMV/total primary infections (IgG positive with IgM positive and low or intermediate avidity).
Neonatal infection rate (congenital CMV) | 6-27 months
  no. PCR-CMV in neonatal urine/total primary infections (IgG positive with IgM positive and low or intermediate avidity).

SECONDARY OUTCOMES:
Congenital CMV sequelae rate at one year of life | 18-36 months
  no. symptomatic cases at one year of life/total primary infections (IgG positive with IgM positive and low or intermediate avidity).
Rate of TOP after diagnosis of primary infections: | 2-19 months
  no. TOP before amniocentesis among cases of primary infection/total primary infection (IgG positive with IgM positive and low or intermediate avidity).
Rate of legal termination of pregnancy after diagnosis of fetal infection | 3-19 months
  no. TOP after positive PCR-CMV in amniotic fluid and no fetal involvement/total primoinfections (IgG positive with IgM positive and low or intermediate avidity).
Rate of TOP after diagnosis of fetal anomalies | 3-19 months
  no. TOP after PCR-CMV in positive amniotic fluid and with fetal involvement/total primoinfections (IgG positive with IgM positive and low or intermediate avidity).
no. TOP after PCR-CMV in positive amniotic fluid and with fetal involvement/total primoinfections (IgG positive with IgM positive and low or intermediate avidity). | 2-18 months
  total number of serologies performed in the 4 centers / number of first visits <14 weeks in the four centers
Annual cost of CMV screening in the first trimester | month 19-24

CONTACTS AND LOCATIONS:
Locations (1):
- ASSIR Metropolitana Nord, Badalona, Spain

IPD SHARING:
Plan to Share IPD: Undecided